CLINICAL TRIAL: NCT07213609
Title: A Phase 1/2 Open-label, Multicenter Study of Oral GSK5460025 Alone or in Combination With Other Anti-cancer Agents in Adult Participants With Mismatch Repair-deficient (dMMR) or Microsatellite Instability-High (MSI-H) Solid Tumors
Brief Title: A Study to Investigate the Safety and Preliminary Efficacy of GSK5460025 Alone or in Combination With Other Anti-cancer Agents in Participants With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 224035; 2025-522318-21 (EudraCT Number)
Record Dates: First submitted 2025-07-04; First posted 2025-10-09 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Neoplasms, Colorectal; Neoplasms
Keywords: GSK5460025; Solid tumors; Colon cancer; Rectal cancer; Colorectal cancer; Endometrial cancer; Mismatch repair deficient; dMMR; microsatellite instability high; MSI-H
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Endometrial Neoplasms; Turcot syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose escalation of GSK5460025 monotherapy (Experimental): Participants will receive GSK5460025 as monotherapy.
  Interventions: Drug: GSK5460025
- Part 2: Dose expansion of GSK5460025 monotherapy (Experimental): Participants will receive GSK5460025 as monotherapy.
  Interventions: Drug: GSK5460025

INTERVENTIONS:
Drug: GSK5460025 — GSK5460025 will be administered

SUMMARY:
Solid tumours are abnormal lumps of tissue that can occur in different parts of the body. The tumours involved in this study have specific genetic characteristics that can make them more aggressive and challenging to treat. The study will test whether GSK5460025 alone or in combination (potential combinations may be included in future amendments to the protocol) with other anti-cancer agents can decrease tumor size, is safe, well-tolerated, and how the drug is processed in the body over time.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically diagnosed advanced (unresectable, metastatic or recurrent) solid tumor
* Has a known dMMR/MSI-H status as determined by a certified local laboratory at the time of Pre-screening or has an unknown Mismatch repair (MMR)/ Microsatellite Instability (MSI) status at the time of Pre-screening and MMR/MSI status will be determined by central reference laboratory
* Provides an archival or fresh (preferred) formalin fixed, paraffin embedded (FFPE) sample
* Intends to receive GSK5460025 as next treatment
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Is expected to have a minimum of 3 months life expectancy
* Has adequate organ function, as defined in the protocol

Part 1 inclusion criteria:

• Has histologically diagnosed advanced (unresectable, metastatic or recurrent) solid tumor and has exhausted all standard of care treatment options

Part 2 inclusion criteria:

* Has histologically diagnosed advanced (unresectable, metastatic or recurrent) Colorectal cancer (CRC) or Endometrial cancer (EC)
* Has received at least 1 but no more than 3 lines of systemic anticancer therapy for their advanced (unresectable, metastatic or recurrent) disease including at least one line of Immune checkpoint inhibitors (ICI) therapy
* Has measurable disease (i.e., at least 1 target lesion) during the Screening period per RECIST 1.1, as determined by the investigator

Exclusion Criteria:

* Has not recovered (i.e., to Grade ≤1 or to baseline) from prior anticancer therapy-induced Adverse Events (AEs)
* Has received prior treatment with a Werner (WRN) inhibitor or Nucleotide Excision Repair Targeting (NERT) agent.
* Is unable to swallow and retain orally administered study treatment
* Has untreated or progressed metastases in brain or CNS
* Has a known additional malignancy that progressed or required active treatment within the last 2 years because reoccurrence of another malignancy would confound interpretation by RECIST 1.1 criteria. Exceptions include basal or squamous cell carcinomas of the skin or in situ carcinomas [e.g., breast, cervix, bladder] that have been resected with no evidence of metastatic disease.
* Has any impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs
* Has cirrhosis or current unstable liver or biliary disease
* Has known hypersensitivity to any of the study interventions or any of their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2028-09-28 (Estimated); Study Completion 2028-10-27 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with dose limiting toxicities (DLTs) per dose level | Up to 28 days
Part 1: Number of participants with treatment emergent serious adverse events (TESAEs) and treatment emergent adverse events (TEAEs) by severity per dose level | Up to approximately 33 months
Part 1: Number of participants with TESAEs and TEAEs by severity per dose level during DLT observation period | Up to 28 days
Part 1: Number of participants with dosage modifications due to TEAEs per dose level | Up to approximately 33 months
Part 2: Objective Response Rate (ORR) | Up to approximately 33 months
  ORR is defined as percentage of participants with confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) by investigator assessment.

SECONDARY OUTCOMES:
Part 1: Plasma concentrations for GSK5460025 | Up to approximately 36 months
Part 1: Area under the concentration-time curve (AUC) for GSK5460025 | Up to approximately 36 months
Part 1: Maximum concentration (Cmax) for GSK5460025 | Up to approximately 36 months
Part 1: Time to maximum concentration (Tmax) for GSK5460025 | Up to approximately 36 months
Part 1: Number of participants with clinically important changes in laboratory parameters, Electrocardiogram (ECGs), and vital signs per dose level | Up to approximately 36 months
Part 2: Number of participants with TESAEs and TEAEs by severity | Up to approximately 36 months
Part 2: Number of participants with TEAEs leading to dosage modifications | Up to approximately 36 months
Part 2: Number of participants with clinically important changes in laboratory parameters, ECGs, and vital signs | Up to approximately 36 months
Part 2: Progression-free Survival (PFS) | Up to approximately 36 months
  PFS is defined as time from first dose to progressive disease (as assessed per RECIST 1.1 by Investigator assessment) or death from any cause, whichever is earlier
Part 2: Duration of Response (DoR) | Up to approximately 36 months
  DoR is defined as time from first documented PR or CR to progressive disease (as assessed per RECIST 1.1 by investigator assessment) or death from any cause, whichever is earlier for participants who have achieved a confirmed CR or PR.
Part 2: Plasma concentration of GSK5460025 | Up to approximately 36 months

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf